CLINICAL TRIAL: NCT04831957
Title: Hypothyroidism After the TAVI Procedure in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nathalie compté, Clinic head of geriatric unit, Universitair Ziekenhuis Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UZCompte3
Record Dates: First submitted 2021-03-19; First posted 2021-04-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Hypothyroidism; TAVI
Keywords: Hypothyroidism; TAVI
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Intervention Model Description: Academic trial, prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient underwent TAVI procedure (Other): - Elderly patients who will undergo a TAVI procedure coming to the geriatric day hospital
  Interventions: Diagnostic Test: Assesment of thyroïd function

INTERVENTIONS:
Diagnostic Test: Assesment of thyroïd function — Blood sample for TSH, fT4, fT3, anti TPO, anti TG thyroid ultra sound Iodine urine sample

SUMMARY:
Aortic stenosis is highly prevalent in advancing age. The prognosis of this disease has dramatically changed with the surgical replacement of the aortic valve and the trans catheter aortic valve re-placement (TAVI). The TAVI procedure is also successful in octogenarians and frail patients. However, the evaluation before the TAVI procedure requires a high dosage of iodinated contrast agent with, consequently, an increased risk for thyroid dysfunction. The primary endpoint of this study is to assess, prospectively, the incidence and the predictive factors (underlying thyroid disease, medication, food preservative, topical antiseptics) of hypothyroidism after a TAVI procedure. The secondary endpoint is the influence of the occurrence of hypothyroidism after the TAVI procedure on the geriatric assessment.

DETAILED DESCRIPTION:
Aortic stenosis is highly prevalent in advancing age. The prevalence is 2.5% at an age of 75 years and 8.1% at an age of 85 years. The estimated mortality after onset of symptoms (dizziness, syncope, thoracic pain and dyspnea) with conventional medical treatment is 75% after 3 years follow up. The prognosis of this disease has dramatically changed with the surgical replacement of the aortic valve. However, an open surgical procedure is not always possible in high risk patients for anatomical reasons (sternotomy, radiation and chest deformation) or comorbidities defined by the Euroscore and the Society of Thoracic Surgeons' risk score (STS score).

Trans-catheter aortic valve replacement (TAVI) is becoming the standard care of patients suffering of non-operable, high risk severe and symptomatic aortic stenosis. The TAVI procedure is associated with immediate hemodynamic improvement characterized by a decreased aortic valve mean pressure gradient, an improved left ventricular end systolic volume and mass, a decreased end ventricular diastolic volume and a better ejection fraction. This hemodynamic improvement translates into better clinical outcomes. Mortality rates (2.2% and 6.7% at one month and at one year) and long term stroke rate are similar after TAVI or surgical replacement.

The TAVI procedure is also successful in octogenarian and in frail patients. Consequently, patient's frailty is a growing argument to refer the patient for a percutaneous treatment of valve disease instead of a conventional surgical approach.

The standard evaluation before the TAVI procedure comprises some radiologic studies with iodinated contrast agent (coronarography, thoracic CT scanner and the TAVI procedure itself). Furthermore, some patients require a treatment with Amiodarone® because of the occurrence of atrial fibrillation during the procedure.

A typical iodinated contrast study confers 13500 µg of free iodine and 15-60g of bound iodine (several hundred thousand times above the recommended daily intake). An excess of iodium expo-sure can lead to thyroid dysfunction:

* Hyperthyroidism particularly in patients with underlying nodular thyroid disease (Jod-Basedow effect).
* Hypothyroidism in patients with underlying thyroid disease or in patients who are taking medication (lithium, amiodarone) which can lead to thyroid dysfunction. The mechanism of iodinated contrast agent hypothyroidism is the failure to escape of the acute Wolf-Chaikoff effect.

Amiodarone confers 3-21 mg iodine daily and can also lead to thyroid dysfunction particularly in patients with underlying thyroid disease because of the failure to escape of the acute Wolf-Chaikoff effect. An autoimmune mechanism is also described.

Epidemiology In our recent clinical practice (geriatric day hospital UZ Brussel), an increased incidence of hypothyroidism in elderly patients after a TAVI procedure has been observed. In our knowledge, there are no data about the incidence of hypothyroidism and what could be the impact for elderly patients after a TAVI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written Informed Consent prior to any study specific proce-dures
* Patient: males and females must be ≥ 70 years old
* Patients who will undergo a TAVI procedure

Exclusion Criteria:

* - No obtained signed, dated and written Informed Consent.
* Known thyroid dysfunction (for example: Basedow, Hashimoto,...)
* Patients receiving any of the following: Lithium, Strumazol or a recent treatment of radio-Iode

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
to assess prospectively the incidence of hypothyroidism after a TAVI procedure. | Baseline, at 4-8-12 weeks
  Change is value of TSH and fT4,
To assess the underlying thyroid disease | At baseline
  Presence of thyroid nodule door ultra sound
To assess the influence of iodinated constrast on hypothyroidism | At 4 weeks
  Value of presence of Iodine in urine sample
To assess the influence of autoimmune disease on hypothyroidism after TAVI | Baseline
  Anti TPO
To assess the influence of presence of antibodies on hypothyroidism after TAVI | Baseline
  Anti TG

SECONDARY OUTCOMES:
to assess the influence of the occurrence of hypothyroidism after the TAVI procedure on dependence level | Baseline and at 1 month
  Value of dependance through :
  - Katz scale (ADL: assessment of activities of daily living): It rates 6 tasks of daily liv-ing (bathing, dressing, toilet, transfer, continence and eating) on a scale from 1 to 4. A low score means absence of dependence, and a high score the maximum of de-pendence for the task
to assess the influence of the occurrence of hypothyroidism after the TAVI procedure on the cognitive function | Baseline and at 1 month
  Value of MMSE (Mini Mental Status Examination): a 0-30 score of cognitive func-tions,<25/30 meaning cognitive function impairment
to assess the influence of the occurrence of hypothyroidism after the TAVI procedure on depression | Baseline and at 1 month
  Value of GDS (geriatric depression scale) a 0-15 score. A score > 15 means risk for depression
to assess the influence of the occurrence of hypothyroidism after the TAVI procedure on mobility | Baseline and at 1 month
  Value of mobility through
  * Tinetti : a 0-28 score : a score < 26 means mobility problems
  * Timed up and go : Impaired mobility if > 12.5s
  * 4 meter walking speed : risico for sarcopenia if speed > 0.7m/s
to assess the influence of the occurrence of hypothyroidism after the TAVI procedure on instrumental daily living | Baseline and at 1 month
  - lawton scale (assessment of instrumentary assessment of activities of daily living) a 0-27 score; a high score means independence; a low score means dependence

CONTACTS AND LOCATIONS:
Locations (1):
- UZ brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
no sharing plan

REFERENCES:
- [Background] Stone ML, Kern JA, Sade RM. Transcatheter aortic valve replacement: clinical aspects and ethical considerations. Ann Thorac Surg. 2012 Dec;94(6):1791-5. doi: 10.1016/j.athoracsur.2012.09.047. No abstract available. PMID 23176901
- [Background] Leontyev S, Walther T, Borger MA, Lehmann S, Funkat AK, Rastan A, Kempfert J, Falk V, Mohr FW. Aortic valve replacement in octogenarians: utility of risk stratification with EuroSCORE. Ann Thorac Surg. 2009 May;87(5):1440-5. doi: 10.1016/j.athoracsur.2009.01.057. PMID 19379882
- [Background] Kodali SK, Williams MR, Smith CR, Svensson LG, Webb JG, Makkar RR, Fontana GP, Dewey TM, Thourani VH, Pichard AD, Fischbein M, Szeto WY, Lim S, Greason KL, Teirstein PS, Malaisrie SC, Douglas PS, Hahn RT, Whisenant B, Zajarias A, Wang D, Akin JJ, Anderson WN, Leon MB; PARTNER Trial Investigators. Two-year outcomes after transcatheter or surgical aortic-valve replacement. N Engl J Med. 2012 May 3;366(18):1686-95. doi: 10.1056/NEJMoa1200384. Epub 2012 Mar 26. PMID 22443479
- [Background] Leung AM, Braverman LE. Iodine-induced thyroid dysfunction. Curr Opin Endocrinol Diabetes Obes. 2012 Oct;19(5):414-9. doi: 10.1097/MED.0b013e3283565bb2. PMID 22820214
- [Background] Trohman RG, Sharma PS, McAninch EA, Bianco AC. Amiodarone and thyroid physiology, pathophysiology, diagnosis and management. Trends Cardiovasc Med. 2019 Jul;29(5):285-295. doi: 10.1016/j.tcm.2018.09.005. Epub 2018 Sep 20. PMID 30309693